CLINICAL TRIAL: NCT05528991
Title: Oxford Classification and Clinical Remission After Initial Treatments in Patients With IgA Nephropathy：a Cohort Study
Brief Title: Oxford Classification and Clinical Remission After Initial Treatments in Patients With IgA Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20223357009
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; Oxford Classification; clinical remission rate
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- mesangial hypercellularity, M: the histopathology was graded based on the revised Oxford Classification system as follows: M absent (M0) or M present (M1)
- endocapillary hypercellularity, E: E absent (E0) or E present (E1)
- segmental glomerulosclerosis, S: S absent (S0) or S present (S1)
- tubular atrophy/interstitial fibrosis, T: T ≤ 25% (T0) or T 26%-50% (T1), or T > 50% (T2)
- crescents, C: C absent (C0) or C present ≥ 1 glomerulus (C1) or C > 25% glomeruli (C2)

SUMMARY:
IgA nephropathy (IgAN) is the most common form of primary glomerulonephritis and one of the leading causes of end-stage renal disease in China. The clinical manifestations of IgAN varies widely among individuals, and renal pathology is crucial for determining the severity of renal damage and predicting the renal progression. However, the association between renal pathology and patient response to medication has not been reported, and the majority of earlier RCT studies have not taken renal pathology into consideration when enrolling patients. The Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group, one of the most prestigious kidney disease organizations in the world, claims that there is not enough evidence to support the use of Oxford Classification to decide whether to administer immunosuppressive therapy to patients with IgAN.Therefore, the goal of this study was to investigate the relationship between Oxford Classification and clinical remission rates following initial teatments in patients with IgAN, with the aim of providing a basis for individualized clinical treatment plans. This study was a single-center prospective cohort study, and patients who were hospitalized in Shenzhen Second People's Hospital from January 2011 to January 2021 and diagnosed as IgAN by renal biopsy were collected continuously and followed up until December 2022. Cox regression models were used to analyze the effect of different Oxford Classifications on the clinical remission rates of patients at 6, 12, 18, and 24 months of treatments, and the relationship between Oxford Classification and secondary outcome indicators such as long-term renal function and urinary protein changes were analyzed using generalized additive mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years；
* Initial renal biopsy；
* Glomeruli>8；
* eGFR>15ml/min；
* Proteinuria/creatinine ratio（PCR）>0.5g/g

Exclusion Criteria:

* Secondary IgAN
* Combined with other kidney diseases
* Combined with acute kidney injury
* Combined with tumor
* Followed-up time <6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Shenzhen Second People's Hospital from January 2011 to January 2021 with IgAN confirmed by renal biopsy were included.
Sampling Method: Non-Probability Sample
Enrollment: 474 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rates (including complete and partial clinical remission rates) at 6, 12, 18, and 24 months for IgAN patients with different Oxford pathology scores (M, E, S, T, C) after being treated with the initial treatments. | 6, 12, 18, and 24 months after being treated with the initial treatments.
  Complete clinical remission: 24h urine protein <0.2g/d (or total urine protein/urine creatinine <0.2g/g) .
  Partial clinical remission: ≥50% decrease in urine protein from baseline and urine protein <1g/d (or total urine protein/urine creatinine <1g/g).

SECONDARY OUTCOMES:
The longitudinal changes in renal function and urinary protein in IgAN patients with different Oxford Classification scores (M, E, S, T, C) after the initial treatments. | During the follow-up period, the study will be terminated if the patient is transferred to renal transplantation, hemodialysis, peritoneal dialysis, or other centers, and the remaining patients will be followed until December 31, 2022
  The rate of change in renal function: the estimated rate of change in glomerular filtration rate (eGFR).
  The rate of change of urine protein: the rate of change of total urine protein/urine creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Wan, Study Director — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 year after publication

REFERENCES:
- [Background] Trimarchi H, Barratt J, Cattran DC, Cook HT, Coppo R, Haas M, Liu ZH, Roberts IS, Yuzawa Y, Zhang H, Feehally J; IgAN Classification Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Conference Participants. Oxford Classification of IgA nephropathy 2016: an update from the IgA Nephropathy Classification Working Group. Kidney Int. 2017 May;91(5):1014-1021. doi: 10.1016/j.kint.2017.02.003. Epub 2017 Mar 22. PMID 28341274
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Coppo R. Towards a personalized treatment for IgA nephropathy considering pathology and pathogenesis. Nephrol Dial Transplant. 2019 Nov 1;34(11):1832-1838. doi: 10.1093/ndt/gfy338. PMID 30476257
- [Background] Lv J, Zhang H, Wong MG, Jardine MJ, Hladunewich M, Jha V, Monaghan H, Zhao M, Barbour S, Reich H, Cattran D, Glassock R, Levin A, Wheeler D, Woodward M, Billot L, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Wang HY, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):432-442. doi: 10.1001/jama.2017.9362. PMID 28763548